CLINICAL TRIAL: NCT01338454
Title: Can we Use Intravenous Injection of Tranexamic Acid in Routine Practice With Active Management of the Third Stage of Labor?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, medical doctor, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: gungorduk12
Record Dates: First submitted 2011-04-11; First posted 2011-04-19 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Obstetrical Hemorrhage
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- tranexamic acid (Active Comparator): TA administered intravenously over a 5 min period at delivery of the anterior shoulder
  Interventions: Drug: transamin
- saline (No Intervention): 10 mL of saline was administered intravenously over a 5 min period at delivery of the anterior shoulder

INTERVENTIONS:
Drug: transamin — TA was administered intravenously over a 5 min period at delivery of the anterior shoulder
  Arms: tranexamic acid

SUMMARY:
Obstetrical hemorrhage accounts for nearly one quarter of all maternal deaths worldwide and was the most common cause of maternal death in the Turkey [1,2]. Most of these deaths occur within 4 h of delivery and are a result of problems during third and fourth stages of labor. It also contributes significantly to serious maternal morbidity. Obstetric, surgical and radiological interventions play central role in the management of obstetric hemorrhage; however, pharmacologic management and in particular prohemostatic therapies also play an important role in the final maternal outcome. Administration of tranexamic acid (TA), intravenously in the third stage of labor may be one of these methods.

TA a synthetic derivate of the amino acid lysine, is an antifibrinolytic that reversibly inhibits the activation of plasminogen, thus inhibiting fibrinolysis and reducing bleeding. TA may enhance the effectiveness of the patient's own hemostatic mechanism [3,4]. In nonobstetric surgery, a systematic review of randomized controlled trails showed that tranexamic acid reduced the risk of blood transfusion [ relative risk (RR) 0.61; 95% CI 0.54-0.69] and also reduced the need for re-operation as a result of bleeding (RR 0.67; 95% CI 0.41-1.09). There was no evidence for an increased risk of thrombotic events [5].

In gynecology and obstetrics, TA is most commonly used to treat idiopathic menorrhagia, and is an effective and well-tolerated treatment when administered orally [5,6,7]. Bleeding associated with pregnancy (placental abruption, placenta previa) has also been treated with TA [6]. Furthermore, four randomized controlled studies have shown that TA reduces postpartum hemorrhage (PPH) following cesarean delivery [7-11]. Only one randomized trail is available evaluating the effect of TA use to prevent bleeding in the postpartum period following spontaneous vaginal delivery [12].

The purpose of our study was to estimate the effect of the addition of intravenous TA to a standard active management of the third stage of labor (which includes prophylactic injection of 10 IU of oxytocin within two minutes of birth, early clamping of the umbilical cord, and controlled cord traction).

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 37 and 42 weeks,
* live fetus,
* cephalic presentation,
* vaginal birth.
* Patients who had a risk factors for PPH, such as multiple gestation, polyhydramnios, fetal macrosomia, antepartum hemorrhage, anemia (haemoglobin concentration < 8 g/dL), severe pre-eclampsia, or coagulopathy

Exclusion Criteria:

* placenta previa,
* placental abruption,
* cesarean section or any uterine scar, abnormal placentation (accreta, increta, or percreta),
* a current or previous history of significant disease, including heart disease, liver, renal disorders.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The amount of blood loss in the third and fourth stages (the fourth stage of labor begins with delivery of the placenta and ends 2 hours after delivery) of labor. | 2 hours
  The volume of blood loss was measured by weighing a sheet soaked from the end of the delivery to 2h after birth. We used a specially designed operating sheet and an electronic scale to weigh all the material (with a 1 g deviation range). The quantity of blood (ml) = (weight of used materials - weight of materials prior to use)/1.05.

SECONDARY OUTCOMES:
incidences of PPH >500 ml | 2 hours
  The quantity of blood (ml) = (weight of used materials - weight of materials prior to use)/1.05 > 500 mL
the incidences of severe postpartum hemorrhage | 2 hours
  The quantity of blood (ml) = (weight of used materials - weight of materials prior to use)/1.05 ≥1000 ml
need for additional uterotonic drugs | 2 hours
  need for additional uterotonic drugs such as 200 µg intravenous metylergometrine, 20 IU oxytocin infusion in 500 ml ringer lactate, and/or 800 misoprostol rectally for vaginal bleeding
side effects at time of TA injection | 2 hours
  nausea, vomiting or diarrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Bakıryok Women and Children Hospital, Istanbul, Bakırkoy, Turkey (Türkiye)

REFERENCES:
- [Derived] Gungorduk K, Asicioglu O, Yildirim G, Ark C, Tekirdag AI, Besimoglu B. Can intravenous injection of tranexamic acid be used in routine practice with active management of the third stage of labor in vaginal delivery? A randomized controlled study. Am J Perinatol. 2013 May;30(5):407-13. doi: 10.1055/s-0032-1326986. Epub 2012 Sep 21. PMID 23023559